CLINICAL TRIAL: NCT00462657
Title: Early Diagnosis of Invasive Aspergillosis in a High Risk Group of Patients Using Serum and Bronchoalveolar Lavage Fluid Real Time PCR and Galactomannan ELISA
Brief Title: Early Diagnosis of Aspergillosis in Patients at High Risk of Fungal Infection Caused by Treatment for Hematologic Cancer or Other Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Bartholomew's Hospital (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Diagnostic
Other Study IDs: CDR0000539539; BARTS-PECT2005; EU-20719; PFIZER-BARTS-PECT2005; SPRI-BARTS-PECT2005; GILEAD-BARTS-PECT2005; BARTS-05/Q0603/68
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2007-09

CONDITIONS: Graft Versus Host Disease; Infection; Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: infection; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; de novo myelodysplastic syndromes; myelodysplastic/myeloproliferative neoplasm, unclassifiable; previously treated myelodysplastic syndromes; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; graft versus host disease
MeSH Terms: conditions — Graft vs Host Disease; Infections; Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Congenital Abnormalities; Myeloproliferative Disorders; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — Polymerase Chain Reaction; Bronchoalveolar Lavage; Immunoenzyme Techniques; Bronchoscopy

INTERVENTIONS:
Genetic: polymerase chain reaction
Other: bronchoalveolar lavage
Other: immunoenzyme technique
Other: laboratory biomarker analysis
Procedure: bronchoscopy
Procedure: management of therapy complications

SUMMARY:
RATIONALE: Studying ways to diagnose fungal infections early may help doctors plan the best treatment.

PURPOSE: This clinical trial is studying laboratory tests to see how well they find aspergillosis early in patients at high risk of fungal infection caused by treatment for hematologic cancer or other disease.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the test characteristics of galactomannan (GM) ELISA using serum and bronchoalveolar lavage fluid (BALF) collected from patients at high risk of invasive fungal infection.
* Determine the test characteristics of aspergillus PCR using blood and BALF samples collected from these patients.
* Evaluate the role of noninvasive exhaled breath condensate (EBC) in detecting invasive aspergillosis (IA).
* Determine whether repeated measures over time or a combination of markers improves the test characteristics.
* Establish cutoff points for the diagnosis of IA.

Secondary

* Determine the inflammatory marker and cytokine profile of EBC in fungal infection and after bone marrow transplantation as a marker of acute lung injury.
* Assess the role of bronchoscopy with bronchoalveolar lavage in identifying the causal pathogen early in the disease course of febrile neutropenic patients.
* Assess the role of GM ELISA in prognosis and response to treatment for IA.
* Assess the role of aspergillus PCR in prognosis and response to treatment for IA.

OUTLINE: This is a prospective study.

Patients are assessed for early diagnosis of invasive aspergillosis (IA) using serum and bronchoalveolar lavage fluid (BALF) evaluated by ELISA for galactomannan (GM) antigen and real time PCR for fungal DNA. Serum samples are collected at baseline and periodically during study, beginning with the onset of neutropenia and continuing until resolution of fever or recovery of neutrophil count. BALF samples are collected in patients with abnormal chest radiology evaluated by bronchoscopy and bronchoalveolar lavage. BALF is analyzed for GM antigen, fungal DNA, inflammatory markers, and cytokines.

Patients are also assessed using exhaled breath condensate (EBC) evaluated by GM ELISA and real time PCR. EBC is collected at baseline and periodically during study to detect GM antigen or fungal DNA and to measure markers of pulmonary inflammation and oxidative stress (e.g., pH, hydrogen peroxide, and leukotriene B4).

PROJECTED ACCRUAL: A total of 200 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* At high risk for developing invasive aspergillosis (IA) due to any of the following risk factors:

  * Diagnosis of acute myeloid leukemia, myelodysplastic syndromes, or acute lymphoblastic leukemia AND meets ≥ 1 of the following criteria:

    * Receiving intensive chemotherapy with expected duration of neutropenia (ANC < 500/mm³) of > 10 days
    * Receiving high-dose steroids
  * Concurrent treatment with allogeneic hematopoietic stem cell transplantation (HSCT)
  * Requirement for high-dose steroids for graft-versus-host disease after HSCT
  * History of probable or proven IA and receiving chemotherapy
* No preexisting chest disease

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2005-07

PRIMARY OUTCOMES:
Sensitivity and specificity of galactomannan (GM) ELISA and real time PCR in detecting invasive aspergillosis (IA)
Diagnostic value of IA screening by GM ELISA and real time PCR, in terms of positive and negative predicative values

CONTACTS AND LOCATIONS:
Overall Officials: Samir G Agrawal, MD, PhD, Study Chair — St. Bartholomew's Hospital
Locations (2):
- United Kingdom (2):
  - Saint Bartholomew's Hospital, London, England
  - Royal Brompton Hospital, London, England